CLINICAL TRIAL: NCT01417429
Title: Galantamine Effects on Nicotine Responses in Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mehmet Sofuoglu, Mehmet Sofuoglu, M.D.,Ph.d., Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HIC1001006227; NCT01417429 (Registry Identifier: Clinical trials)
Record Dates: First submitted 2011-04-05; First posted 2011-08-16 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Smoking; Tobacco Withdrawal
Keywords: galantamine; subjective nicotine; tobacco withdrawal symptoms; nicotine
MeSH Terms: conditions — Smoking | interventions — Galantamine; Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Galantamine (Active Comparator): galantamine will be given with intravenous nicotine
  Interventions: Drug: Galantamine
- Nicotine (Experimental): Subject will be given IV Nicotine
  Interventions: Drug: IV Nicotine

INTERVENTIONS:
Drug: Galantamine — 8mg/a day or placebo
  Other Names: Razadyne, Razadyne ER
  Arms: Galantamine
Drug: IV Nicotine — 1.0 mg/70 kg of nicotine against saline
  Other Names: liquid nicotine
  Arms: Nicotine

SUMMARY:
This will be a 2-4 week double-blind, placebo-controlled study. Twenty four male and female smokers will first have two 4-day treatment periods, in which they will be randomized to galantamine (8 mg/day) or placebo. These treatment periods will be separated by a 3 to 14 day washout period. During the first 3-days of each treatment period, smokers will have daily clinic visits, where they will receive study medications and any adverse effects from study medications will be monitored. Starting at 10 p.m. on Day 1 of each treatment period, subjects will refrain from smoking for approximately 2.5 days, until the experimental session on Day 4. Compliance with non-smoking will be verified by CO levels < 10 ppm. During the experimental sessions, subjects will receive saline or 1.0 mg/70 kg of nicotine intravenously in a random, double-blind manner. The sequence of nicotine treatments will be counterbalanced among subjects such that equal number of subjects will receive saline first or nicotine first. Following each saline and nicotine treatments, physiological, subjective and cognitive measurements will be obtained

DETAILED DESCRIPTION:
In this double-blind, crossover study, the investigators are proposing to evaluate galantamine's effects on the subjective nicotine effects and the severity of tobacco withdrawal symptoms. Twenty four male and female smokers will first have two 4-day treatment periods, in which subjects will be randomized to galantamine (8 mg/day) or placebo. These treatment periods will be separated by a 3 to 14 day washout period. This range of washout period, while minimizing carryover medication effects between treatments, will provide flexibility for subjects to comply with study procedures. During study participation, subjects will be instructed to continue to smoke as usual during the study except the 2.5 days of smoking abstinence before each test session. Starting at 10 p.m. on Day 1 of each treatment period, subjects will refrain from smoking for approximately 2.5 days, until the test session on Day 4. Subjects will have twice daily outpatient visits during the first 3 days and a test session on day 4. During the outpatient visits, study medication will be administered and tobacco withdrawal symptoms and compliance with smoking abstinence will be monitored. On Day 4 of each treatment phase subjects will have a test session, where they will receive saline or 1.0 mg/70 kg of nicotine intravenously in a random, double-blind manner. The sequence of nicotine treatments will be counterbalanced among subjects such that equal number of subjects will receive saline first or nicotine first. Following each saline and nicotine administration, physiological, subjective and cognitive measurements will be obtained.

Currently 12 subjects completed this protocol. This study is in data analysis. (April 2011)

ELIGIBILITY:
Inclusion criteria:

* female and male smokers, aged 18 to 55 years;
* history of smoking daily for the past 12 months, at least 15 cigarettes daily;
* CO level > 10ppm;
* for women: not pregnant as determined by pregnancy screening, nor breast feeding, and using acceptable birth control methods.

Exclusion criteria:

* history of major medical illnesses including asthma or chronic obstructive lung disease, history or current gastrointestinal ulcer, hepatic or renal impairment and cardiac rhythm disturbances or other medical conditions that the study physician deems contraindicated for the subject to be in the study;
* regular use of psychotropic medication (antidepressants, antipsychotics, or anxiolytics) and/or recent psychiatric diagnosis and treatment for Axis I disorders including major depression, bipolar affective disorder, schizophrenia and panic disorder within the past year;
* current dependence on alcohol or on drugs or treatments for drug or alcohol addiction ;
* use of drugs that slow heart rate (eg, beta-blockers), which may increase the risk of bradycardia and AV block, or NSAIDs, which may increase potential for developing ulcers/active or occult gastrointestinal bleeding;
* known allergy to galantamine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Galantamine Effects on Nicotine Responses in Smokers | 1 year to complete
  Urine sample and blood samples anticipated for 24 male and females

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D., Ph.D., Principal Investigator — Yale University
Locations (1):
- Department of Veterans Affairs, West Haven, Connecticut, United States